## CONSENT FORM: Effectiveness of mHealth and Teach-Back methods in readmissions reduction in Prime Minister's National Health Programme A Feasibility Randomized Controlled Trial

**Dated: 1 Feb 2020** 

## **Part 1: Consent Form**

I am a research student and am working on a research project titled "Effectiveness of m Health and Teach Back methods in readmissions reduction in Prime Minister's National Health Programme – A Feasibility Randomized Controlled Trial".

I need to collect some information from you regarding your admission and comorbidities. I am inviting you to be my study participant and need 15-20 minutes of your time for a face to face interview for information related to this research project.

I might call you later depending on the group you are assigned to if you give consent to participate in the trial.

Take your time and decide whether you want to participate in this interview or not.

This interview does not provide any benefits of any type.

You may refuse to participate at any time even after the interview session has started.

Your identity will be confidential and will not be disclosed to anyone without your permission. I may be using words that you do not comprehend. Please feel free to ask anything and stop me anytime during this information transfer phase.

| Do you wish to particip | ate? | |
|---|---|---|
| Yes | No | |
| Consent by participant | Part 2: Certificate of Consent: | |
| | nation provided to me or the information h | as been read to me. |
| | to participate as participants in this resear | |
| Signature of the Participa | ants: | |
| Date:(d | ay/month/year) | |
| | | Participants |
| Statement by person ta | king consent: | |
| I have correctly read out | t all the information to the potential partic | ipant and to best of my ability |
| made sure that he/she un | derstands that the research process. | |
| Name of the person takir | ng consent: | |
| Signature of the person to | aking consent: | |
| Date: | ( day/month/year) | |